CLINICAL TRIAL: NCT02325583
Title: Baskent University Institutional Review Board
Brief Title: Intraoral 30% Glucose Effect In Newborns
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, H. Evren Eker, Assocciate Professor, Baskent University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KA14/299
Record Dates: First submitted 2014-12-17; First posted 2014-12-25 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Epilepsy; Hydrocephaly
Keywords: Intraoral 30% glucose, newborn, MRI
MeSH Terms: conditions — Epilepsy; Hydrocephalus | interventions — Glucose; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intraoral 30% Glucose in Newborns (Experimental): 0.5-1 mL 30% glucose solution was administered orally and the motionless and sleepiness of newborn was evaluated. If the target conditions was not achieved, 0.5-1 mL increments of glucose was added. After 2 consecutive oral glucose administration the newborns who did not keep motionless or sleep and had motion artefacts sedated with midazolam. The routine blood glucose level measurement was also performed in ICU.
  Interventions: Drug: 30% Glucose; Drug: Midazolam

INTERVENTIONS:
Drug: 30% Glucose — ORAL 30% GLUCOSE 0,5-2 ML
  Other Names: POLİFLEKS %30 DEKSTROZ POLİFARMA İLAÇ 05.10.2014/204-71
Drug: Midazolam — INTRAVENOUS 0.1 MG/KG MIDAZOLAM
  Other Names: ZOLAMİD 5 MG/ML, DEFARMA İLAÇ SAN, 406036

SUMMARY:
Newborn often sedated during MRI but sedation itself creates adverse events and management is more challenging in the MR environment. The investigators describe the investigators initial experience with oral 30% glucose administration through a pacifier during MRI for imaging of newborns. Using this technique, majority of newborns can complete MRI examination without the need for sedation and also offers the availability of administering sedatives to unsuccessful patients.

DETAILED DESCRIPTION:
19 consecutive newborns over 10 months period were assessed retrospectively. 0.5-1 mL 30% glucose solution was administered orally and after suckling, the motionless and sleepiness of newborn was evaluated. If the target conditions was not achieved, 0.5-1 mL increments of glucose was added. After 2 consecutive oral glucose administration the newborns who did not keep motionless or sleep and had motion artefacts sedated with midazolam. The outcome measure was the success of the procedure which was determined by providing qualitative images appropriate for interpretation following 30% glucose administration. The routine blood glucose level measurement of the newborns after imaging procedures in the ICU was also performed for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Newborns admitted from newborn intensive care unit for MR imaging

Exclusion Criteria:

* Intubated newborns

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of newborn provided qualitative images for MRI following oral glucose administration | 10 months

REFERENCES:
- [Background] Skogsdal Y, Eriksson M, Schollin J. Analgesia in newborns given oral glucose. Acta Paediatr. 1997 Feb;86(2):217-20. doi: 10.1111/j.1651-2227.1997.tb08872.x. PMID 9055897